CLINICAL TRIAL: NCT02824523
Title: Role of PDG2 in the Aspirin-Induced Reactions and in the Treatment of Aspirin-Exacerbated Respiratory Disease
Brief Title: Role of Inflammatory Mediators in AERD
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Tanya Laidlaw, MD, Associate Physician, Brigham and Women's Hospital
Other Study IDs: 2016P001164
Record Dates: First submitted 2016-06-24; First posted 2016-07-06 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Asthma, Aspirin-Induced
Keywords: asthma; nasal polyps; aspirin sensitivity; AERD
MeSH Terms: conditions — Asthma, Aspirin-Induced; Asthma; Nasal Polyps | interventions — Aspirin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- High-dose aspirin
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: aspirin

SUMMARY:
The purpose of this research study is to learn new information about the underlying cause of aspirin-exacerbated respiratory disease (AERD) and the benefit of high-dose aspirin therapy. AERD is a disease that involves asthma, recurring nasal polyps, and respiratory reactions to aspirin and other nonsteroidal anti-inflammatory drugs. This study will be conducted on individuals with AERD who are referred to the Brigham and Women's Hospital AERD Center for clinical evaluation and potential aspirin desensitization. Desensitization to aspirin and subsequent treatment with daily high-dose oral aspirin is standard of care for patients with AERD who do not respond adequately to steroids and have recurrent nasal polyposis or symptomatic asthma. This study will involve five visits to Brigham and Women's Hospital and will align closely with the standard of care for the treatment of AERD.

ELIGIBILITY:
Inclusion Criteria:

* History of asthma
* History of nasal polyposis
* History of at least one clinical reaction to oral aspirin or other nonselective COX inhibitor with features of both lower (cough, chest tightness, wheezing, dyspnea) and upper (rhinorrhea, sneezing, nasal obstruction, conjunctival itching and discharge) airway involvement
* Stable asthma (post-bronchodilator FEV1 of ≥70%, no use of oral or systemic steroids for at least 1 month, and no hospitalizations or emergency room visits for asthma for the prior 6 months) at the time of entry into the study
* Currently taking montelukast as part of standard asthma treatment for at least 4 weeks before the V1 visit

Exclusion criteria:

* Pregnancy or current breastfeeding
* History of bleeding diathesis or use of anticoagulant or antiplatelet drugs
* History of thrombocytopenia < 50 x 10^9/L
* Hypersensitivity to montelukast
* Peptic ulcer disease
* Unstable asthma (post-bronchodilator FEV1 of less than 70%, use of oral or systemic steroids for at least 1 month prior to visit 1, or hospitalizations or emergency room visits for asthma for the prior 6 months)
* Use of zileuton (which can mask symptoms of aspirin-induced reaction) within 1 month prior to the V1 visit
* Age under 18 or over 75 years
* Current smoking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aspirin-exacerbated respiratory disease who are undergoing aspirin desensitization and starting high-dose aspirin therapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Therapeutic efficacy of high-dose aspirin as assessed by asthma symptom control (Asthma Control Questionnaire) | 8 weeks
Therapeutic efficacy of high-dose aspirin as assessed by change in lung function | 8 weeks
Therapeutic efficacy of high-dose aspirin as assessed by change in sinus symptoms (Sino-Nasal Outcome Test) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tanya M Laidlaw, MD, Principal Investigator — Brigham and Women's Hospital; Katherine C Cahill, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Patel PP, Cui J, Cahill KN, Laidlaw TM. Objective validity of patient-reported symptoms in aspirin-exacerbated respiratory disease patients. Clin Exp Allergy. 2022 Feb;52(2):348-351. doi: 10.1111/cea.14062. Epub 2021 Dec 1. No abstract available. PMID 34820927
- [Derived] Staso PJ, Wu P, Laidlaw TM, Cahill KN. Scoring tool for systemic symptoms during aspirin challenge detects mediator production in aspirin-exacerbated respiratory disease. Ann Allergy Asthma Immunol. 2021 Jul;127(1):131-133. doi: 10.1016/j.anai.2021.03.025. Epub 2021 Mar 27. No abstract available. PMID 33781934